CLINICAL TRIAL: NCT00980304
Title: A Multicenter, Open Label, Phase II Trial of Rituximab in Combination With ICE as Salvage Therapy in the Relapsed DLBCL Patients After 1st Line Induction Treatment of 6-8 Cycles of RCHOP-LIKE Chemo
Brief Title: R Retreatment in 1st Relapsed DLBCL
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Shen, Zhixiang / Professor, Ruijin Hospital Affiliated to Shanghai JiaoTong University School of Medicine
Other Study IDs: ML22515
Record Dates: First submitted 2009-09-18; First posted 2009-09-21 (Estimated); Last update posted 2009-09-21 (Estimated); Status verified 2009-09

CONDITIONS: Lymphomas
Keywords: Diffuse large B cell lymphomas
MeSH Terms: conditions — Lymphoma; Dendritic Cell Sarcoma, Interdigitating | interventions — Rituximab

ARMS (1):
- Rituximab in combination with ICE as salvage therapy (Experimental)
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Rituximab

SUMMARY:
It is a phase II , multicenter, open label clinical trial. Only the relapsed DLBCL patients after 1st line induction treatment of 6~8 cycles of RCHOP-like chemo will be enrolled to receive 3 cycles of RICE as salvage therapy.

After treatment each patient should be followed up for 2 years.

ELIGIBILITY:
Inclusion Criteria:

1. Relapsed DLBCL patients having received 6 - 8 cycles of RCHOP-like chemotherapy as 1st line induction treatment.
2. Disease relapsed no earlier than 6 months after prior induction treatment.
3. Confirmed CD20 positivity of the lymphoma at time of diagnosis (prior to induction therapy)
4. ECOG performance status of 0, 1 or 2 at time of inclusion (see Appendix IV )
5. Known IPI at time of diagnosis (prior to induction therapy)
6. Age ≥18 years and <65 y
7. Life expectancy of > 3 months
8. Be willing and able to comply with the protocol for the duration of the study
9. Agree to use effective contraception for the entire treatment period and during the 12 months thereafter
10. Patient's written informed consent

Exclusion Criteria:

1. More than one prior chemoimmunotherapy regimen.
2. Histologies other than DLBCL according to the WHO/REAL classification
3. History of malignancy other than squamous cell carcinoma, basal cell carcinoma of the skin, surgically treated malignant melanoma or carcinoma in situ of the cervix within the last 5 years.
4. Major surgery, other than diagnostic surgery, within the last 4 weeks.
5. Evidence of CNS involvement patients
6. Unacceptable hematologic status at baseline prior to study start below any of the values listed: WBC: <3 x 109/L; absolute neutrophil count (segmented + bands) <1.5 x 109/L; platelets: <100 x109/L
7. Abnormal liver function tests prior to study start above any of the values listed: serum bilirubin >2 mg/dL (30 mmol/L); ALAT or ASAT >2.5 x upper limit of normal range; or Abnormal renal function (serum creatinine > 150 μmol/L ).
8. HIV-positive patients.
9. Contraindication to the investigational medication
10. Active viral hepatitis, specifically HBV or HCV infection
11. Serious underlying medical conditions, (e.g. ongoing infection, uncontrolled diabetes mellitus, severe cardiac dysfunction or angina, gastric ulcers, active autoimmune disease)
12. Life expectancy < 3 months
13. Treatment within a clinical trial within 30 days prior to trial entry
14. Women who are breast feeding, are not using effective contraception, are pregnant
15. Patients under tutelage

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult